CLINICAL TRIAL: NCT00933816
Title: Phase I/II Study of Sorafenib In Combination With Low-dose FP Intraarterial Infusion Chemotherapy
Brief Title: Study of Sorafenib In Combination With Low-dose 5-fluorouracil/Cisplatin (FP) Intraarterial Infusion Chemotherapy
Acronym: SILIUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kindai University (Other)
Responsible Party: Japan Liver Oncology Group, Japan Liver Oncology Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JLOG0901
Record Dates: First submitted 2009-07-01; First posted 2009-07-07 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: sorafenib; intraarterial infusion chemotherapy; Low dose FP; cisplatin; fluorouracil
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib with Low-dose FP (Experimental)
  Interventions: Drug: sorafenib, cisplatin, fluorouracil

INTERVENTIONS:
Drug: sorafenib, cisplatin, fluorouracil — Sorafenib will be administered orally at a dose of 400 mg bid for 28 days in the all patients. Cisplatin at the dose of 10-20 mg/m2 will be administered at day 1 and day8, and fluorouracil at the dose of 170-330 mg/m2 will be administered continuously at day 1-day 5, and day8-day12 via the implanted catheter system. A cycle is defined as 28 days and 3 cycles of this combination therapy will be continued.
  Other Names: sorafenib with hepatic arterial infusion of low dose FP

SUMMARY:
The purpose of this study is to determine the recommended dose of the combination therapy of sorafenib with hepatic arterial infusion of low dose cisplatin and fluorouracil on patients with advanced hepatocellular carcinoma (Phase I), and to evaluate the efficacy of this combination therapy in the recommended dose (Phase II).

DETAILED DESCRIPTION:
In Phase I, there will be 9 to 18 patients enrolled. Cohorts of 3 to 6 patients will receive escalated dose of cisplatin and fluorouracil until the MTD is reached. There will be no intra-patient dose escalation. Sorafenib will be administered orally at a dose of 400mg bid for 28 days in the all patients. Cisplatin at the dose of 10-20mg/m2 will be administered at day 1 and day8, and fluorouracil at the dose of 170-330mg/m2 will be administered continuously at day1-day5, and day8-day12 via the implanted catheter system. A cycle is defined as 28 days and 3 cycles of this combination therapy will be continued. At the end of each cycle, adverse effect will be evaluated and dose escalation will be determined. In Phase II, there will be 28 patients enrolled. Time to progression of this combination therapy at the recommended dose will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. 20 Years and older.
2. Life expectancy of at least 12 weeks at the pre-treatment evaluation.
3. Advanced hepatocellular carcinoma with histological evidence on a biopsy specimen, or typical findings by dynamic CT or CT during hepatic arteriography/arterioportography.
4. Not suitable for resection or local ablation therapy or transcatheter arterial chemoembolization.
5. One treatment of hepatic arterial infusion chemotherapy without implanted catheter system is allowed.
6. ECOG Performance status of 0 or 1.
7. Cirrhotic status of Child-Pugh class A or B.
8. Adequate bone marrow, liver and renal function, as assessed by the following laboratory requirements:

   * Hemoglobin 8.5 g/dl
   * Granulocytes 1500/μL
   * Platelet count 50,000 /μL
   * PT-INR 2.3 or PT 6 seconds above control
   * Total serum bilirubin 2 mg/dl
   * AST(SGOT) and ALT(SGPT) 5 × upper limit of normal
   * Serum creatinine 1.5 × upper limit of normal
   * Amylase 5 × upper limit of normal
9. Written Informed Consent must be obtained.

Exclusion Criteria:

1. Previous malignancy (except for cervical carcinoma in situ, adequate treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis and T1], early gastric cancer, or other malignancies curatively treated > 3 years prior to entry
2. Renal failure
3. Any heart disease as follows

   * Congestive heart failure defined as NYHA class III or IV
   * Active coronary artery disease or ischemic heart disease such as cardiac infarction within 6 months prior to screening
   * Serious cardiac arrhythmia
   * Serious hypertension
4. Active clinically serious infections.
5. Active chicken pox.
6. Auditory disorder.
7. Known history of HIV infection.
8. Known metastatic or meningeal tumors.
9. Extrahepatic tumor spread.
10. History of seizure disorder.
11. Clinically significant gastrointestinal bleeding within 4 weeks prior to study entry.
12. Embolization or infarction such as transient ischemic disease, deep vein thrombosis, pulmonary embolization).
13. Any history of treatment as follows:

    * Treatment with the agent which induces CYP3A4
    * Surgical procedure within 4 weeks prior to start of study drug
    * History of organ allograft
14. Patients unable to swallow oral medications.
15. Gastrointestinal disease that may affect to the absorption of drug or pharmacokinetics.
16. Medication that may affect to the absorption of drug or pharmacokinetics.
17. Any disease or disorder that may affect the evaluation of study drug.
18. Entry to the other clinical trial within 4 weeks prior to entry to this study.
19. Pregnant or breast-feeding patients.
20. Known allergy to the investigational agent or any agent given in association with this trial.
21. Substance abuse, medical, psychological or social conditions that, in the judgment of the investigator, is likely to interfere with the patient's participation in the study or evaluation of the stuy results.
22. Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity in phase I and Time to progression in Phase II | Every 4 weeks

SECONDARY OUTCOMES:
Phase I and II: Overall survival (OS) | Every day
Phase I and II: Progression free survival (PFS) | Every four weeks
Phase I: Time to progression (TTP) | Every four weeks
Phase I and II: Response Rate (RR) | Every four weeks
Phase I and II: Adverse effect (AE) | Every four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masatoshi Kudo, Principal Investigator — Kindai University
Locations (3):
- Japan (3):
  - Kurume University Medical Center, Kurume, Fukuoka
  - Ogaki Municipal Hospital, Oogaki, Gifu
  - Kinki University School of Medicine, Ōsaka-sayama, Osaka